CLINICAL TRIAL: NCT03891264
Title: Investigation of Cannabidiol for Reduction of NeuroInflammation in Chronic Back Pain
Acronym: CBD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding obtained to do a larger placebo-controlled trial
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jodi Gilman, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019P000852
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Back Pain, Low
MeSH Terms: conditions — Low Back Pain | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CBD Arm (Experimental): Evaluation with Magnetic Resonance-Positron Emission Tomography Imaging and/or behavioral pain assessment before and after a 4-week trial of a liquid formulation of CBD.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Epidiolex, an agent within the anti-epileptic drug class, will be used. Epidiolex, Greenwich Biosciences Inc.'s CBD formulation, is a 100 mg/mL purified oral solution. The recommended starting dosage is 2.5mg/kg taken twice daily (5mg/kg/day). After one week, the dosage will be increased to a maintenance dosage of 10 mg/kg twice daily (20 mg/kg/day). At the end of the first week, the patient will increase the dose to 10 mg/kg twice daily for the following week.
  Other Names: Epidiolex

SUMMARY:
In this research, the study team will use brain imaging to evaluate the presence of neuroinflammation in the brains and spinal cords of patients with low back pain, and whether CBD effects levels of neuroinflammation. The efficacy of CBD use for low back pain treatment will also be evaluated by observing whether CBD administration will reduce neuroinflammation and low back pain symptoms.

DETAILED DESCRIPTION:
The goal of this research study is to test whether "glial cells" (the immune cells of the brain and spinal cord) that are active in patients with low back pain can be reduced with CBD. Previous studies have showed that patients with chronic low back pain demonstrated elevations in brain levels of the 18kDa translocator protein (TSPO), a marker of glial activation.

To test this hypothesis, the study team will image the brains and spinal cords of patients suffering from low back pain using integrated magnetic resonance- positron emission tomography (MR-PET), and a radiotracer called [11C]PBR28, which tracks levels of glial activation.

The efficacy of CBD as a treatment for chronic low back pain will be evaluated. The study team will observe whether 4 weeks of CBD treatment may reduce glial activation along with self-reported low back pain symptoms. To this end, patients will be evaluated clinically and/or re-scanned after completing the 4-week trial of minocycline.

This study will be enrolling individuals who have been suffering from chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 and ≤ 75;
* the ability to give written, informed consent;
* ongoing pain that averaged at least 4, on a 0-10 scale of pain during a typical week, and present for at least 50% of days during a typical week;
* fluency in English;
* on a stable pain treatment (pharmacological or otherwise) for the previous four weeks.
* Medical records confirming diagnosis of low back pain
* Chronic low back pain, ongoing for at least 6 months prior to enrollment.

Exclusion Criteria:

* outpatient surgery within 2 months and inpatient surgery within 6 months from the time of scanning;
* elevated baseline transaminase (ALT and AST) levels above 3 times the Upper Limit of Normal (ULN), accompanied by elevations in bilirubin above 2 times the ULN
* any interventional pain procedures within 6 weeks prior to scanning procedure or at any point during study enrollment;
* surgical intervention or introduction/change in opioid regimen at any point during study enrollment
* contraindications to functional magnetic resonance imaging scanning and positron emission tomography scanning (including presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia);
* current or past history within the last 5 years of major medical illness not affecting the central nervous system, other than chronic pain;
* implanted spinal cord stimulator (SCS) for pain treatment;
* any history of neurological illness or major medical illness affecting the central nervous system, unless clearly resolved without long-term consequences;
* current or past history of major psychiatric illness;
* PTSD, depression, and anxiety are exclusion criteria only if the conditions were so severe as to require hospitalization in the past year.
* pregnancy or breast feeding;
* history of head trauma requiring hospitalization;
* major cardiac event within the past 10 years;
* any use of recreational drugs in the past 3 months
* any marijuana use, medical or recreational, in the past 3 months
* an abnormal physical exam (e.g., peripheral edema);
* routine use of opioids ≥ 60 mg morphine equivalents;
* use of immunosuppressive medications, such as prednisone, TNF medications within 2 weeks of the visit;
* current bacterial or viral infection;
* Any other contraindications to CBD administration noted by the study physician.
* If undergoing blood draws through an arterial line during scan, contraindications to placement of arterial line, such as abnormal result on modified Allen's test on both hands; Raynaud syndrome; bleeding disorder; use of anticoagulants such as Coumadin, Plavix or Lovenox

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Gilman, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make this data available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after 2 years
Access Criteria: Researchers, not for commercial use

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBD Arm
Started | 7
Received Intervention | 3
Completed | 2
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | CBD Arm
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Positron Emission Tomography Signal
Description: The investigators will test for the presence of a significant treatment effect in the brain [11C]PBR28 signal.
Time Frame: 4 weeks
Population: Trial ended early because funding was obtained to do a larger, placebo-controlled trial.
Measure: Mean (Standard Deviation); unit: Standardized Uptake Values (SUVs)
Arm/Group | CBD Arm
Number analyzed (Participants) | 2
Standardized Uptake Values (SUVs) | 0.00197 (0.017756865)

2. Secondary Outcome: Changes in Pain Outcomes as Measured by Self Report on a 0-10 Numerical Pain Rating Scale (Worst Pain in the Past 24 Hours).
Description: The investigators will test for the presence of a significant treatment effect in pain outcomes on a self reported numerical (0-10) pain rating scale. Higher number indicates worse pain.
Time Frame: 4 weeks
Population: Trial ended early because funding was obtained to do a larger, placebo-controlled trial.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBD Arm
Number analyzed (Participants) | 2
score on a scale | 4.5 (0.707106781)

ADVERSE EVENTS:
Time Frame: From enrollment to 2 weeks following study medication discontinuation (6 weeks)
Arm/Group | CBD Arm
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBD Arm (N=3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03891264/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03891264/ICF_001.pdf